CLINICAL TRIAL: NCT06660992
Title: Phase 3 Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of HSK31858 in Participants With Non-cystic Fibrosis Bronchiectasis
Brief Title: A Study to Assess the Efficacy and Safety of HSK31858 in Participants With Non-Cystic Fibrosis Bronchiectasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK31858-301
Record Dates: First submitted 2024-09-23; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK31858 40mg (Experimental): HSK31858 40mg treat for 52-week
  Interventions: Drug: HSK31858, tablet
- Placebo (Placebo Comparator): the placebo comparator of study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK31858, tablet — HSK31858 is a novel inhibitor of DPP1 developed by Hisco Pharmaceutical and can reduce pulmonary exacerbations over a 52-week treatment period in patients with non-cystic fibrosis bronchiectasis
  Arms: HSK31858 40mg
Drug: Placebo — the placebo comparator of study
  Arms: Placebo

SUMMARY:
This is a phase III, randomized, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of HSK31858 in non-cystic fibrosis bronchiectasis (NCFBE) participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years and BMI≥18.0 kg/m^2 at the time of signing the ICF. 2. Chest HRCT showed bronchiectasis affecting one or more lobes and was confirmed by a clinician as NCFBE(clinically characterized by chronic cough, expectoration and/or intermittent hemoptysis, with or without shortness of breath and respiratory failure). HRCT was considered effective if the patient had received HRCT in the same hospital within 12 months and screening HRCT is not necessary.

  3. Have at least 2 pulmonary exacerbations in the past 12 months before Screening.

  4. If long-term treatment with bronchodilators (long-acting β-agonists and/or long-acting muscarinic antagonists) is required, the dose and regimen should remain stable for at least 3 months before the screening visit and throughout the study period.

  5. The estimated survival time ≥ 12 months. 6. Women must be post-menopausal, surgically sterile, or using highly effective contraception methods from Day 1 to at least 30 days after the last dose.

  7. Males with female partners of childbearing potential must be using effective contraception from Day 1 to at least 90 days after the last dose.

  8. Give their signed study informed consent to participate.

Exclusion Criteria:

* 1. Have a primary diagnosis of COPD or asthma as judged by the Investigator. 2. A history of malignancy (excluding cured basal cell carcinoma of the skin, carcinoma in situ, and papillary carcinoma of the thyroid gland. The patients who had survived lung cancer surgery for at least 5 years without antitumor therapy can enroll in the study ) within 5 years prior to screening or a history of antitumor therapy.

  3. Have bronchiectasis due to CF (HRCT showed that the above lung diseases became predominant) as judged by the Investigator.

  4. Currently being treated Non-tuberculous Mycobacterial (NTM) pulmonary infections, allergic bronchopulmonary aspergillosis, or tuberculosis (TB), or active and currently symptomatic infections caused by COVID-19, or have the history of bronchopulmonary aspergillosis.

  5. Patients with severe pulmonary fibrosis such as lung destruction, pneumonectomy surgery history, and pneumoconiosis, as well as previous or existing decompensated stage of pulmonary heart disease.

  6. Patients who had experienced any degree of acute exacerbation of bronchiectasis or were developing an acute exacerbation of bronchiectasis before 4 weeks of screening.

  7. Patients who had hemoptysis and required medical intervention within 4 weeks prior to screening(except for coughing up minorbloody streaks).

  8. Patients previously treated with HSK31858 or other DPP1 inhibitor products. 9. Subjects with uncontrolled hypertension (SBP ≥180 mmHg at rest and/or DBP ≥110 mmHg). 10. Subjects with uncontrolled type 1 or type 2 diabetes (fasting plasma glucose >7.0 mmol/L).

  11. Subjects with a history of liver disease or current treatment for liver disease during the screening period, including but not limited to acute or chronic hepatitis, cirrhosis or liver failure (except for mild to moderate non-alcoholic fatty liver disease).

  12. Active hepatitis B virus infection (hepatitis B surface antigen positive with HBV-DNA load above the lower limit of detection), active hepatitis C virus infection (HCV antibody positive with HCV-RNA load above the lower limit of detection), or known HIV infection or syphilis infection.

  13. Any other unstable clinical condition, including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematologic, psychiatric, or major physiological dysfunction, that the investigator considers to be (a) likely to affect patient safety throughout the study; (b) Influence the results of the study and its interpretation; (c) impeding the patient's ability to complete the entire study.

  14. Laboratory tests during the screening period meet the following conditions:
  1. AST>2.0×ULN or ALT>2.0×ULN or TBIL>1.5×ULN
  2. eGFR<60ml/min/1.73m2
  3. Hb<90 g/L
  4. WBC <3×109 /L
  5. PLT <70×109 /L
  6. INR>1.5ULN，PT>ULN+3s, or APTT>ULN+10s. 15. Had participated in a clinical trial of any other drug or medical device in the 3 months prior to the screening (a drug or medical device treated with a clinical trial) or the subject had not been more than 5 half-lives from the last clinical trial of the drug at the time of screening.

     16. Medications that may cause hyperkeratosis (e.g., tumor necrosis factor-α antagonists) within 4 weeks prior to screening.

     17. Patients who have used a strong inducer or suppressor of CYP3A within 14 days or 5 half-lives of the first investigational drug (whichever is longer).

     18. Patients who had smoked an average of 10 cigarettes or more per day in the previous 1 year were screened.

     19. Pregnancy and lactation. 20. The subjects were unable to complete the questionnaires due to their limited educational level, or the subjects and their families failed to fill in the subjects' log cards.

     21. Had received live attenuated vaccine within 30 days before randomization. 22. The investigators judged that there were other conditions that were not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
Frequency of pulmonary exacerbations | week 52

SECONDARY OUTCOMES:
Time to first pulmonary exacerbation | week 52
Change from Baseline(Screening) in forced expiratory volume in 1 second (FEV1) | week 52
Change from Baseline(Screening) in 24-hour Sputum Weight and Sputum purulence score | week 52
  score from 0 to 8
Change from Baseline in the Respiratory Symptoms Domain Score of the Quality of Life (QOL) Bronchiectasis questionnaire | week 52
  score from 0 to 100

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Yixing People's Hospital, Yixingcun, Jiangxi

IPD SHARING:
Plan to Share IPD: Undecided